CLINICAL TRIAL: NCT05533801
Title: An Open-Label, Parallel-Group, Randomized Study to Demonstrate the Bioequivalence of the Subcutaneous Formulation of Lecanemab Supplied in Vials and a Single-Use Auto-Injector
Brief Title: A Study to Demonstrate the Bioequivalence of Lecanemab Supplied in Vials and a Single-Use Auto-Injector (AI) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BAN2401-A001-005
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: BAN2401; Lecanemab
MeSH Terms: interventions — lecanemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: Lecanemab 720 mg (Experimental): Participants will receive a single SC dose of lecanemab 720 milligram (mg) in the lower abdomen using a vial and syringe on Day 1.
  Interventions: Drug: Lecanemab
- Treatment B: Lecanemab 720 mg (Experimental): Participants will receive a single SC dose of lecanemab 720 mg in the lower abdomen using AI on Day 1.
  Interventions: Drug: Lecanemab

INTERVENTIONS:
Drug: Lecanemab — Lecanemab will be administered subcutaneously using a vial and syringe.
  Other Names: BAN2401
  Arms: Treatment A: Lecanemab 720 mg
Drug: Lecanemab — Lecanemab will be administered subcutaneously using AI.
  Other Names: BAN2401
  Arms: Treatment B: Lecanemab 720 mg

SUMMARY:
The primary purpose of this study is to demonstrate the bioequivalence (BE) of a single subcutaneous (SC) dose of lecanemab via vial and AI in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, male or female, age greater than or equal to (>=) 18 years and less than or equal to (<=) 65 years at the time of informed consent. To be considered non-smokers, participants must have discontinued smoking for at least 4 weeks before dosing
2. Body Mass Index >=18 and less than (<) 30 kilogram per square meter (kg/m^2) at Screening

Exclusion Criteria:

1. Clinically significant illness that requires medical treatment within 8 weeks of dosing or a clinically significant infection that requires medical treatment within 4 weeks of dosing
2. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; example, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
3. Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5 half-lives of the other investigational drug, whichever is longer, preceding informed consent
4. Prior exposure to lecanemab, or any other anti-amyloid therapies
5. Hypersensitivity to lecanemab or any of the excipients, or to any (monoclonal anti-body [mAb]) treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
AUC(0-t): Area Under the Serum Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration for Lecanemab | 0 (Pre-dose), 4, 8, 24, 48, 72, 96, 120, 168, 336, 504, 696, 840, 1176 hours post-dose
AUC(0-inf): Area Under the Serum Concentration-time Curve From Time Zero to Time Extrapolated to Infinity for Lecanemab | 0 (Pre-dose), 4, 8, 24, 48, 72, 96, 120, 168, 336, 504, 696, 840, 1176 hours post-dose
Cmax: Maximum Observed Serum Concentration for Lecanemab | 0 (Pre-dose), 4, 8, 24, 48, 72, 96, 120, 168, 336, 504, 696, 840, 1176 hours post-dose
Tmax: Time to Reach the Maximum (Peak) Serum Concentration for Lecanemab | 0 (Pre-dose), 4, 8, 24, 48, 72, 96, 120, 168, 336, 504, 696, 840, 1176 hours post-dose
t1/2: Terminal Elimination Phase Half-life for Lecanemab | 0 (Pre-dose), 4, 8, 24, 48, 72, 96, 120, 168, 336, 504, 696, 840, 1176 hours post-dose

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to Day 50
  A TEAE is defined as an adverse event (AE) that emerges during treatment, having been absent at pretreatment (baseline) or reemerges during treatment, having been present at pretreatment (baseline) but stopped before treatment, or worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
Number of Participants With Abnormal Laboratory Values | Baseline up to Day 22
  Clinical laboratory parameters will include hematology, blood chemistry, and urinalysis.
Number of Participants With Abnormal Vital Signs Values | Baseline up to Day 50
  Vital sign parameters will include diastolic and systolic blood pressure (BP), pulse rate, respiratory rate, body temperature and body weight.
Number of Participants With Anti-drug Antibodies (ADAs) | Baseline up to Day 50
  ADAs will be measured using validated electrochemiluminescent immunoassay methods.
Number of Participants With Neutralizing Antibodies (NAbs) | Baseline up to Day 50
  NAbs will be measured using validated electrochemiluminescent immunoassay methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.